CLINICAL TRIAL: NCT00740571
Title: A Randomised Controlled Trial in the Palliative Setting Regarding Off-Label Medication: Investigating the Efficiency of Amitriptyline Versus Pregabalin From a Societal Perspective
Brief Title: Amitriptyline or Pregabalin to Treat Neuropathic Pain in Incurable Cancer
Acronym: Off-label
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other); University of Amsterdam (Other)
Responsible Party: K.C.P. Vissers MD, PhD, FIPP, Radboud University Nijmegen Medical Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80-82310-98-8612
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Cancer; Neuralgia
Keywords: neuralgia; off-label; cancer
MeSH Terms: conditions — Neoplasms; Neuralgia | interventions — Amitriptyline; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Strategy in which patient starts with amitriptyline
  Interventions: Drug: amitriptyline
- 2 (Active Comparator): Strategy in which patient starts with pregabalin
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: amitriptyline — strategy in which the patient starts with amitriptyline, during 8 weeks
  Other Names: tryptizol
  Arms: 1
Drug: pregabalin — Strategy in which patient starts with pregabalin
  Other Names: lyrica
  Arms: 2

SUMMARY:
Rationale: Often, incurable cancer patients suffer from severe symptoms as (neuropathic) pain and fatigue with polypharmaceutic interventions as a consequence. Regarding neuropathic pain in incurable cancer patients, pregabalin has been registered for neuropathic non-cancer pain, and amitriptyline is not registered for neuropathic pain, but is recommended as the drug of first choice in the Dutch handbooks of palliative care. As a consequence of an adaptation of a Dutch law (July 2007) about off-label medication prescription, off-label medication is not allowed anymore unless a standard or protocol exists. No clinical trials for this patient group have been published before.

Objective: To compare efficacy, side effects and costs of a strategy with amitriptyline as drug of first choice versus a strategy with pregabalin as drug of first choice.

Study design: An open label, randomised non-inferiority trial Study population: Incurable cancer patients with neuropathic pain Intervention: When a patient decides to take part in the study, he will be allocated randomly to one of the two study groups. A minimisation algorithm will be used, that balances for the cause of neuropathic pain (tumour related versus treatment related), type of treatment (ongoing chemo- or radiotherapy versus not ongoing chemo- or radiotherapy) and institution. Each drug will be prescribed in a step up procedure. Patients will be followed during 8 weeks.

Main study parameters/endpoints: Neuropathic pain, as measured with the mean VAS and McGill questionnaire, strategy success, costs per strategy, side effects, quality of life and concomitant analgesic drugs.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are hardly any risks for the patients. The drugs in both arms already are usual care for the target population. If there is no or a too small effect, the drug of the other arm will be added, which strategy also is already usual care. All other medication, except for Tricyclic Antidepressants Drugs (TADs) and Anti Epileptic Drugs (AEDs), as well as radiotherapy and chemotherapy are allowed. The patient has to visit the hospital 2 times during the study period. The patient had to fill in a pain diary daily (5 min), cost diary and EQ-5D every other week (10 min), related questionnaires as HADS, McGill and EORTC-QLQ-C30 monthly (20 min).

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Incurable cancer
* Life expectancy three months or longer
* NRS ≥ 4
* Neuropathic pain
* Adequate renal function with cockroft ≥ 60 ml/min
* Signed informed consent
* Expected adequacy of follow up

Exclusion Criteria:

* Previous use of TAD or AED for neuropathic pain within 30 days prior to screening
* Unstable regime of analgetica for 1 week prior to screening
* Use of cannabis
* Radiotherapy aimed at the source of the neuropathic pain 2 weeks before screening
* Chemotherapy with known neurotoxic effect (taxanes, thalidomide, vinca alkaloids, cytarabine,fluoropyrimidines, oxaliplatin) 2 weeks before screening
* Unstable regime of corticosteroids for 1 week prior to screening
* Pregnancy
* Any condition preventing the intake or absorption of oral drugs
* Participation in any other studies involving investigational products within the 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
VAS score | 8 weeks

SECONDARY OUTCOMES:
EQ-5D, McGill, EORTC-C30, HADS | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kris Vissers, MD PhD FIPP, Study Director — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - VUMC, Amsterdam, North Holland
  - Erasmus MC, Rotterdam, South Holland